CLINICAL TRIAL: NCT00314327
Title: Optimizing Response in Psychosis Study
Acronym: ORP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment for the study was limited.
Sponsor: Northwell Health (Other)
Collaborators: The Zucker Hillside Hospital (Other); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Delbert Robinson, MD, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05.04.161
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Psychotic Disorder Not Otherwise Specified
Keywords: first episode; schizophrenia; risperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- long-acting injectable risperidone (Experimental): One week of oral risperidone dosage started at 2mg for the first day and then increased to 4mg. If no side effects are noted, participants are started on the long-acting risperidone. The usual dosage of long-acting risperidone in the study will be 25mg every 2 weeks for a total of 12 weeks. The medication will be administered intramuscularly via injection.
  Interventions: Drug: long-acting injectable risperidone

INTERVENTIONS:
Drug: long-acting injectable risperidone — One week of oral risperidone dosage started at 2mg for the first day and then increased to 4mg. If no side effects are noted, participants are started on the long-acting risperidone. The usual dosage of long-acting risperidone in the study will be 25mg every 2 weeks for a total of 12 weeks. The medication will be administered intramuscularly via injection.
  Other Names: Risperdal (oral) & Risperdal Consta

SUMMARY:
The purpose of this project is to evaluate the efficacy of long-acting risperidone for patients with first episode schizophrenia spectrum who did not improve sufficiently with the first antipsychotic medication they tried during their initial treatment trial.

DETAILED DESCRIPTION:
The goal of the proposed pilot study is to investigate the feasibility and efficacy of the long-acting injectable form of the second generation antipsychotic, risperidone, for the treatment of first episode patients who fail to respond to 12 weeks of treatment with an oral antipsychotic. The rationale for using this long-acting medication is that it eliminates covert non-adherence, which may be a factor in poor response. In addition, pharmacokinetic and pharmacodynamic differences between injectable and oral formulations may result in differences in treatment response favoring the injectable form. Subjects who have not responded sufficiently to treatment with an antipsychotic will be approached for the proposed long-acting risperidone trial. Risperidone treatment will be open label with titration based upon individual response (within FDA approved dose ranges). Treatment will begin with a phase of supplementation with oral risperidone. Subjects will stop their previous antipsychotic, start 2 mg of oral risperidone per day for one day and then increase the dose to 4 mg per day. Subjects who tolerate one week of oral risperidone will then begin injections of 25 mg long-acting risperidone every 2 weeks for a total of 12 weeks. If clinically indicated, the dose may be increased up to a maximum of 50 mg as per FDA guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-IV-defined diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder, or psychotic disorder NOS as assessed using the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID-I/P) (First et al, 1998)
* Is in the first episode of illness. First episode is defined as having had 6 months or less of lifetime treatment with an antipsychotic.
* Has not responded sufficiently to treatment with an antipsychotic. Lack of response is defined as a rating at study entry of 4 (moderate) or more on at least one of the following BPRS-A items: conceptual disorganization, grandiosity, hallucinatory behavior, unusual thought content.
* Continuous antipsychotic treatment at the time of study entry of a minimum of 12 weeks with the same antipsychotic agent.
* Antipsychotic dosing at some point during the 12 weeks must have reached a sufficient dose for antipsychotic response (e.g. patients who received only low dose quetiapine for insomnia or anxiety would not qualify). Sufficient dose for second generation antipsychotics is defined as a minimum dose of risperidone 3 mg/day, olanzapine 10 mg/day, quetiapine 500 mg/day, ziprasidone 100 mg/day or aripiprazole 15 mg/day. Sufficient dose for first generation antipsychotics is defined as 3 mg/day of haloperidol or its equivalent for other first generation agents.
* Aged 15 to 40.
* If age 18 or older, competent and willing to sign informed consent.
* If under age 18, parent or guardian consent and subject assent.
* For women, a negative urine pregnancy test and agreement to use a medically accepted method of birth control.

Exclusion criteria:

* Meets DSM-IV criteria for a current substance-induced psychotic disorder, a psychotic disorder due to a general medical condition, delusional disorder, brief psychotic disorder, shared psychotic disorder, or a mood disorder (major depression or bipolar) with psychotic features.
* Persistence of psychotic symptoms due to nonadherence to antipsychotic medication.
* Medical contraindications to treatment with long-acting injectable risperidone.
* Serious neurological or endocrine disorder or medical condition /treatment known to affect the brain.
* A medical condition requiring medication with psychotropic effects.
* Clinical assessment that trial participation is contraindicated due to risk for homicidal or suicidal behavior.
* A diagnosis of diabetes (fasting glucose > 126 mg/dl).
* Requires with antidepressant or mood stabilizing medication.
* Previous treatment with a long acting formulation of an antipsychotic

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2006-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Delbert G Robinson, M.D., Principal Investigator — The North Shore-Long Island Jewish Health System
Locations (2):
- United States (2):
  - SUNY Downstate Medical Center, Brooklyn, New York
  - The Zucker Hillside Hospital, Glen Oaks, New York

REFERENCES:
- See also: web site of NARSAD — http://www.narsad.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Long-acting Injectable Risperidone
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Long-acting Injectable Risperidone
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response Based Upon BPRS and CGI Ratings
Time Frame: 13 weeks
Arm/Group | Long-acting Injectable Risperidone
Number analyzed (Participants) | 0

2. Secondary Outcome: Negative Symptoms
Description: Zero patients were analyzed as only one subject consented to the study and dropped out of the study before they were randomized. The negative symptoms that were going to be analyzed include: Affective Flattening, Alogia, Avolition /Apathy, and Anhedonia/Asociality
Time Frame: 13 weeks
Population: Zero patients were analyzed as only one subject consented to the study and dropped out of the study before they were randomized.
Arm/Group | Long-acting Injectable Risperidone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Long-acting Injectable Risperidone
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes